CLINICAL TRIAL: NCT06850389
Title: PMCF Investigation of Medical Device ChitoCare® Medical
Status: Recruiting | Type: Observational
Sponsor: Primex ehf (Industry)
Collaborators: Porta Medica (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHITODERM
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Dermatitis; Acne; Conditions After Dematosurgical Procedures; Scars
MeSH Terms: conditions — Dermatitis; Acne Vulgaris; Cicatrix

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ChitoCare® medical Wound Healing Gel — ChitoCare® medical Wound Healing Gel is a medical device containing ChitoClear® chitosan. The device is indicated for the treatment of acute and chronic wounds and other skin conditions, including partial thickness burn wounds.
Device: ChitoCare® medical Healing Spray — ChitoCare® medical Healing Spray is a medical device containing ChitoClear® chitosan. The device is indicated for the treatment of acute wounds and other skin conditions.

SUMMARY:
This is a post-marketing observational clinical investigation conducted as part of the post-market clinical follow-up of ChitoCare® Medical, aimed to confirm safety and efficacy according to the requirements of Regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017 on medical devices, for the following indications:

Gel - scars, conditions after dermatosurgical procedures, dermatitis, acne

Spray - conditions after dermatosurgical procedures, dermatitis, acne

ELIGIBILITY:
The inclusion criteria are fully according to indications:

* Gel - scars, conditions after dermatosurgical procedures, dermatitis, acne
* Spray - conditions after dermatosurgical procedures, dermatitis, acne

The criteria for exclusion are fully according to contraindications:

* Allergy to any of the ingredients of the product

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The device is intended for use in all age groups, including children and the elderly. All participants who fulfill the inclusion and exclusion criteria will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Significant improvement in Vancouver Scar Scale (VSS) | 3 months
  For scars and conditions after dermatosurgical procedures, efficacy is defined as a significant improvement in Vancouver Scar Scale (VSS) scores from baseline after 3 months of treatment.
Significant improvement in Comprehensive Acne Severity Scale (CASS) | 2 months
  For acne, efficacy is defined as a significant improvement in the severity rating of patients' acne using the Comprehensive Acne Severity Scale (CASS) from baseline after 2 months of treatment.
Significant improvement in dermatitis severity scale | 2 months
  For dermatitis, efficacy is defined as a significant improvement in the severity dermatitis severity scale after 2 months of treatment.

SECONDARY OUTCOMES:
Confirmation of safety (adverse events) | 2-3 months
  Safety will be confirmed when less than 5% of subjects report an adverse event when all participants have completed the trial.
Confirmation of safety (serious adverse events) | 2-3 months
  Safety will be confirmed when less than 1% of subjects report a serious adverse event when all participants have completed the trial.
Quality of life assessment (adults) | 2-3 months
  Quality of life will be assessed in adults using the Dermatology Life Quality Index (DLQI) questionnaire. Improvements in quality of life from baseline will be reported.
Quality of life assessment (children) | 2-3 months
  In children, quality of life will be assessed using the pediatric version of the Dermatology Life Quality Index - the Childhood Dermatology Life Quality Index (CDLQI) questionnaire. Improvements in quality of life from baseline will be reported.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Dermatovenerology department, FN Motol, Prague
  - Dermatology of Prof. Hercogova, Prague

IPD SHARING:
Plan to Share IPD: No